CLINICAL TRIAL: NCT02620618
Title: Intravitreal Infliximab in Refractory Uveitis in Behcet's Disease: A Safety and Efficacy Clinical Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tamer Ahmed Macky, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intravitreal Infliximab
Record Dates: First submitted 2015-11-26; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Behçet's Disease; Uveitis
Keywords: Safety; Efficacy; intravitreal infliximab; ocular behcets; refractory posterior uveitis
MeSH Terms: conditions — Behcet Syndrome; Uveitis; Uveitis, Posterior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravitreal Infliximab (Experimental): Patients with refractory behcets uveitis.
  Interventions: Drug: Intravitreal Infliximab

INTERVENTIONS:
Drug: Intravitreal Infliximab — ocular safety and efficacy in treating inflammation in uveitis patients with Behcets Disease
  Other Names: Intravitreal TNF alpha

SUMMARY:
Intravitreal injection of up to 2 mg of infliximab has proved to be safe in animal models (rabbits and primates). These studies have shown no evidence of intraocular inflammation or toxicity by clinical, electrophysiological, and histopathological examination for up to 90 days even with 3 repeated monthly injections. However, the study conducted by Rassi et al was the only one to report the development of severe intraocular inflammation in one eye out of 12 rabbit eyes at 90 days following 3 intravitreal injections (2mg monthly). Unfortunately, clinical studies conducted on patients, so far, have raised serious concern about its safety and adverse effects.

These clinical studies have shown various and inconsistent results in terms of the safety and efficacy of intravitreal infliximab. These studies were conducted on patients with refractory as well as naïve cases of age related macular degenerations choroidal neovascularization (AMD CNV), diabetic macular edema (DME), central retinal vein occlusion (CRVO), angiomatous malformations, pseudophakic macular edema, and uveitis. The doses used ranged from 0.5mg to 2mg. The initial study by Theodossaidis et al in 2009 did not report any intraocular inflammation in 3 patients receiving 2 intravitreal injections of 1 and 2 mg for refractory AMD CNV with 7 months follow up period.(8) Later several clinical studies have reported severe intraocular inflammation following intravitreal injections of infliximab in non-uveitic patients.These collected data have initiated a call for cautious use of intravitreal infliximab.

On the other hand, studies investigating intravitreal infliximab in uveitis patients have shown improvement in vision, reduction in macular thickness on optical coherence tomography (OCT), and reduction in inflammation. In this study, we have investigated the safety and efficacy of 3 consecutive intravitreal infliximab injections (1 mg/0.05 mL, 6 weeks apart) in carefully selected group of patients with refractory uveitis in Behcet's disease.

DETAILED DESCRIPTION:
Approval of the study was obtained from the hospital's ethical committee. The study design and methodology followed the tenets of Declaration of Helsinki. All patients were provided with written informed consent and received a thorough explanation of the study design, aims, and the off-label use of infliximab, its potential risks, and benefits. This is a prospective non-comparative interventional study. The study was conducted on 20 eyes of 20 patients with refractory posterior uveitis in Behçet's disease who received 3 consecutive intravitreal injections of infliximab (1 mg/0.05 ml) 6 weeks apart. Behçet's diseases was diagnosed based on the International Criteria for Behçet's Disease (ICBD).

Patients were subjected to the following initial examinations: best-corrected visual acuity (BCVA) measurement; slit-Lamp examination; measuring intraocular pressure (IOP) by Goldman applanation tonometry; dilated fundus examination by indirect ophthalmoscope; and slit-lamp biomicroscopy including vitritis grading (0-4) and presence or absence of vasculitis, retinitis and papillopathy. Patients also had the following at baseline: fluorescein angiography (FFA), ERG, and central foveal thickness (CFT) OCT (Stratus III OCT; Carl Zeiss, Dublin, CA). Grading of vitritis was as follows: Grade 0: Good view of NFL (nerve fibre layer), Grade +1: clear optic nerve & vessels but hazy NFL, Grade +2: optic nerve & vessels are hazy, Grade +3: view of optic nerve only, and Grade +4: no optic nerve view.

Follow up clinical examinations were at day 1, and weeks 2, 4, 6, 8, 12 and 18. Each follow up visit included: BCVA, slit-Lamp examination, IOP, dilated fundus examination with grading of vitritis (0-4), and presence or absence of vasculitis, retinitis or papillopathy. CFT OCT, and ERG were done at 4, 12 and 18 weeks. FFA was done at the discretion of the examiner and not at every post-injection evaluation.

The intravitreal dose of infliximab used in this study is 1mg/0.05ml. Animal studies have shown intravitreal infliximab in doses up to 2mg is safe clinically, and by electrophysiological and histopathological examinations. These findings were maintained for 3 months with 3 monthly injections. However, in clinical trial severe intraocular inflammation was elicited with even a single low dose of 0.5mg in non-uveitic eyes. Since the 1 mg dose was shown to be effective in controlling inflammation in one study, we decided to use this dose and avoid the 1.5mg and the 2mg doses.

Drug preparation: A vial containing 100 mg of commercially available infliximab powder (Remicade Janssen Pharmaceutical Egypt) was reconstituted with 5 mL of sterile water, and 0.05 mL of this solution (1mg of infliximab) used for each patient and placed in a tuberculin syringe using aseptic techniques. The remaining syringes will be kept in a sterile package at 2-8ºC for 6 weeks.

Injection technique: The eye was prepared in a standard fashion using 5% povidone-iodine, an eyelids speculum to stabilize the eyelids, and the injection of 1mg (0.05 mL) was performed 3.5mm to 4 mm posterior to the limbus, through the infero-temporal pars plana with a 30-gauge needle under topical anesthesia. After the injection, retinal artery perfusion is checked and patients were instructed to administer topical antibiotics for 3 days. All patients were given detailed post-injection instructions and asked to call promptly if any pain or significant changes in vision occurred.

Patients were seen on follow ups and repeated injections were given at 6 weeks intervals if re-injection criteria were met: 1) No evidence of significant ERG changes, 2) No evidence of adverse effects to the drug, 3) Signs of anatomical and/or functional improvement during the first 6 weeks.

Statistical Analysis: Data were statistically described in terms of mean ± standard deviation (±SD), median and range, or frequencies (number of cases) and percentages when appropriate. Comparison of numerical variables between the study groups was done using Freidman's test with Conover test for paired (matched) samples as posthoc multiple 2-group comparisons. For comparing categorical data, Chi square (±2) and McNemar tests were performed. GCC was done using McNemar test. Agreement was tested using kappa statistic. Correlation between various variables was done using Spearman rank correlation equation. P values less than 0.05 was considered statistically significant. All statistical calculations were done using computer program SPSS (Statistical Package for the Social Science; SPSS Inc., Chicago, IL, USA) version 15 for Microsoft Windows Stats Direct statistical software version 2.7.2 for MS Windows, StatsDirect Ltd., Cheshire, UK.

ELIGIBILITY:
Inclusion criteria:

Refractory posterior uveitis in patients with Behçet's disease.

Exclusion criteria:

1. Patients receiving or who had received systemic infliximab or other TNFα inhibitors
2. Patients with uncontrolled systemic Behçet
3. Patients who received previous intravitreal steroids (< 6 months)
4. Patients with severe media opacity
5. Patients with previous history of ocular surgery other than cataract surgery
6. Cataract surgery within the previous 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity in logMAR | 18 weeks
Central Foveal Thickness in microns by Optical Coherence Tomography | 18 weeks
Electroretinogram a and b waves amplitudes in microvolts | 18 weeks
Vitritis severity graded 0-3 | 18 weeks
Electroretinogram a and b waves implicit times in milliseconds | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Soliman, MD PhD, Study Chair — Cairo University